CLINICAL TRIAL: NCT01446757
Title: Effectiveness of a Comprehensive CGA on Frailty in Community-dwelling Elderly People - A Randomised, Controlled Trial
Brief Title: Ambulatory Geriatric Evaluation - Frailty Intervention Trial
Acronym: AGE-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Swedish Association of Local Authorities and Regions (Other)
Responsible Party: Principal Investigator, Anne Ekdahl, Senior Consultant, geriatrician, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011/41-31
Record Dates: First submitted 2011-09-19; First posted 2011-10-05 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Frail Elderly; Deaths
Keywords: quality of life; feeling of security; costs; multiprofessional team; geriatric competence
MeSH Terms: conditions — Death | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The intervention group (Experimental): The intervention group will receive Comprehensive Geriatric Assessment and follow up as a complement to the same standard health care services as the control group. The Comprehensive Geriatric Assessment and follow up will be provides through an outpatient facility that tailors care from a holistic perspective and, based on each patient's individual needs in line with the policy program that Sweden's pensioners' organizations have presented in 2010 together with the Swedish Association of Geriatric Medicine. The team includes, among other things. a. geriatricians, nurses, physiotherapists, assistance officer, dietician, pharmacist and co-operation with the dental hygienist.
  Interventions: Procedure: The intervention group
- Control group (Placebo Comparator): The control group will receive care in the same way as usual meaning access to primary care, hospital in- and outpatient care and care received by the municipality. The only difference between the two groups are that the control group will not have access to the geriatric care team.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: The intervention group — Medical assessment (co-morbid condition, physical and neurological examination, medication review, nutrition, and blood-tests to identify anaemia, diabetes, metabolism and liver- and kidney function); assessment of functioning (ADL/IADL, fall risk), psychological assessment (cognitive decline and depression) and assessment of social and environmental conditions. The care plan is based on the CGA and will be individualised and carried out in discussion with the patient and his/her caregivers. The care will be carried out by an inter-professional Geriatric Team with employees from both the county council and the municipality. The team consists of a core team (including geriatrician and nurse) and a support team (including a social worker, occupational therapist, dietician, pharmacist, physiotherapist, and dental hygienist). The care will involve treatment for unstable medical conditions and support of patients and their caregivers. The team will have regular team conferences.
  Other Names: Geriatric care team
  Arms: The intervention group
Procedure: control group — No intervention
  Arms: Control group

SUMMARY:
The main purpose of this randomised controlled trial is to study if a Comprehensive Geriatric Assessment (CGA) and follow up for community-dwelling elderly people can improve outcomes such as health and health-related quality of life among both patients and relatives, feeling of safety among both patients and relatives and reduce costs, compared with usual care.

DETAILED DESCRIPTION:
Frail older adults are at increased risk of vulnerability and serious health problems. This leads to increased suffering and higher healthcare utilization. There are major gaps in the knowledge needed to create the most favourable care model for preventing frailty and increasing health-related of life. The purpose of this randomised controlled trial is to study if a Comprehensive Geriatric Assessment and follow up in community-dwelling elderly people can prevent frailty, hospitalisation and adverse effects of frailty, improve health and health-related quality of life, and reduce costs, compared with usual care. In a randomized, controlled trial with 24 months of follow-up, a total of 430 older adults with multimorbidity will be randomized into two groups. The intervention group will receive Comprehensive Geriatric Assessment and follow up and the same standard health care services as the control group. The Comprehensive Geriatric Assessment and follow up will be provides through an outpatient facility that tailors care from a holistic perspective and, based on each patient's individual needs in line with the policy program that Sweden's pensioners' organizations have presented in 2010 together with the Swedish Association of Geriatric Medicine. The team includes, among other things. a. geriatricians, nurses, physiotherapists, assistance officer, dietician, pharmacist and co-operation with the dental hygienist.

The primary outcome is development of frailty and hospitalization. Secondary outcomes are adverse effects of frailty, health and health-related quality of life and costs. There is a knowledge gap of how health care can identify persons with frailty and risks for frailty and how to meet their specific care needs. The study aims to fill a clinically important knowledge gap that can guide further development of future care for older people with multi-morbidity and frailty. CGA is readily transferable to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Elderly 75 years and above
* Have been hospitalized three or more times in the last 12 months
* Have three or more diagnoses in their medical records according to the International Classification of Diseases (ICD-10)
* Live in their own homes (not nursing home) in the municipality of Norrkoeping
* Accept to participate in the study.

Exclusion criteria:

- Fulfilling the inclusion criteria but living in a special accommodation for the elderly

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 383 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Hospitalisation | 24 months
  Number of hospitalisations and in-care stays during the trial
Frailty | 24 months
  Unintentional weight loss ≥5% of the previous year. Exhaustion is assessed by two questions from the Centre for Epidemiologic Studies-Depression Scale. Low physical activity includes assessment of habitual physical activity level by using the Swedish version of the International Physical Activity Questionnaire short version (IPAQ-S).Slow walking speed is determined from the better of two attempts at usual "comfortable" walking speed over 4 m with or without a walking aid. Weakness (muscle strength) is assessed by maximal grip strength.

SECONDARY OUTCOMES:
Cognition | 0 and 24 months
  Cognition is assessed by the Mini-Mental State Examination
Symptoms | 0 and 24 months
  Symptoms experienced during the previous week (frequency, intensity, and distress) are assessed by the "The Memorial Symptom Assessment Scale" (MSAS), which measures 32 different symptoms.
Depression | 0 and 24 months
  Depression is assessed using the Geriatric Depression Scale (GDS-15
Health related quality of life | 0 and 24 months
  Health related quality of life (HRQL) is assessed by using the Nottingham Health Profile, first part (NHP) and the generic "EuroQol" questionnaire (EQ-5D)
Nutrition | 0 and 24 months
  The Mini Nutritional Assessment form (MNA), is used to assess nutritional status. The MNA includes 18 items.
Activities of Daily Living | 0 and 24 months
  Barthels index
Falls | 0 and 24 months
  the patient is asked about falls in the last 6 months
Costs | 24 months
  1) Contact and extent of contact with the municipality measured by working hours 2) Number of: visits to day-care centres, in-hospital stays (type of clinic and extent of these), visits to primary care facilities, geriatric ambulatories or other specialist ambulatories 3) Admissions to nursing care facilities
Feeling of security of the patient | 0, 12 and 24 months
  Questionnaire
Feeling of security of the relatives | 0, 12 and 24 months
  Questionnaire
Quality of life of relatives | 0, 12 and 24 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anne W Ekdahl, Physisian, Principal Investigator — Linkopeing University
Locations (1):
- Department of Geriatric Medicine, Norrköping, Sweden

REFERENCES:
- [Derived] Klompstra L, Ekdahl AW, Krevers B, Milberg A, Eckerblad J. Factors related to health-related quality of life in older people with multimorbidity and high health care consumption over a two-year period. BMC Geriatr. 2019 Jul 5;19(1):187. doi: 10.1186/s12877-019-1194-z. PMID 31277674
- [Derived] Lundqvist M, Alwin J, Henriksson M, Husberg M, Carlsson P, Ekdahl AW. Cost-effectiveness of comprehensive geriatric assessment at an ambulatory geriatric unit based on the AGe-FIT trial. BMC Geriatr. 2018 Jan 31;18(1):32. doi: 10.1186/s12877-017-0703-1. PMID 29386007
- [Derived] Ekdahl AW, Wirehn AB, Alwin J, Jaarsma T, Unosson M, Husberg M, Eckerblad J, Milberg A, Krevers B, Carlsson P. Costs and Effects of an Ambulatory Geriatric Unit (the AGe-FIT Study): A Randomized Controlled Trial. J Am Med Dir Assoc. 2015 Jun 1;16(6):497-503. doi: 10.1016/j.jamda.2015.01.074. Epub 2015 Feb 18. PMID 25703450